CLINICAL TRIAL: NCT03963284
Title: Evaluation of the Incidence of Renal Stress by Measuring the NephroCheck Test After Pediatric Cardiac Surgery
Brief Title: Evaluation of AKI by Measuring the NephroCheck Test After Pediatric Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: SCMC/bMX-2019-01
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Acute Kidney Injury; Cardiac Disease; Surgery
MeSH Terms: conditions — Acute Kidney Injury; Heart Diseases | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Procedure: cardiac surgery — pediatric cardiac surgery with cardiopulmonary bypass
Device: NephroCheck test — Urine of the subjects undergoing cardiac surgery with CPB will be tested by NephroCheck test

SUMMARY:
Blood and urine samples of over 200 pediatric subjects (over 28 days to 3 years) undergoing complex cardiac surgery with cardiopulmonary bypass (CPB) will be collected at several time points to measure corresponding biomarkers such as serum creatinine, serum urea concentration, or NephroCheck test ([TIMP-2]*[IGFBP7) to evaluate the diagnostic performance of AKI by NephroCheck test .

DETAILED DESCRIPTION:
At least 200 subjects having undergone pediatric cardiac surgery with cardiopulmonary bypass (CPB). Enrollment will continue with a maximum of 350 subjects until 30 cases of AKI (stage 2 and 3) are reached.

Blood and urines samples will be collected at several time points to measure biomarkers and set up a biobank.

The samples used within the scope of this protocol will be fresh urine samples (1 to 2 ml) and blood samples.

Urine samples for [TIMP-2]*[IGFBP7] measurements will be taken from each subject included in the study during the first 48 hours following cardiopulmonary bypass initiation according to the following schedule:

* baseline before initiation of cardiopulmonary bypass (CPB, 0h).
* - 2h, 4h, 6h, 8h, 12h, 24h, 48h after initiation of CPB

Blood samples for serum creatinine and urea concentration measurement will be taken from each subject included in the study during the first 48 hours following cardiopulmonary bypass initiation according to the following schedule:

* baseline before initiation of cardiopulmonary bypass (CPB, 0h).
* 12h, 24h, 48h, 60h after initiation of CPB

Primary objective:

To evaluate the proportion of subjects predicted to be at risk of AKI (stage 2 and 3) using at least one measurement of NephroCheck in subjects having undergone pediatric cardiac surgery.

Secondary objectives:

* To evaluate the incidence of AKI (stage 2 and 3) according to the KDIGO guideline
* To study the kinetic profile of cell cycle arrest biomarkers (TIMP-2*IGFBP-7) during the first 48 hours in subjects having undergone pediatric cardiac surgery
* To determine the baseline values of [TIMP-2]*[IGFBP7] in the targeted population before surgery
* To determine profile differences of [TIMP-2]*[IGFBP7] between AKI (stage 2 and 3) and non-AKI groups
* To evaluate the diagnostic performances of [TIMP-2]*[IGFBP7] to predict AKI after pediatric cardiac surgery using a cut-off value of 0.3

ELIGIBILITY:
Inclusion Criteria:

* Must sign the consent form
* Clinical diagnosis of complex congenital heart surgery (Risk Adjusted classification for Congenital Heart Surgery [RACHS] score >=2)
* Must undergo elective cardiac surgery with CPB

Exclusion Criteria:

* Clinical diagnosis of severe pre-existing renal insufficiency (SCr >2 times age-adjusted normal range)
* Significant abnormalities of the kidneys or genitourinary tract

Ages: 28 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: At least 200 subjects having undergone pediatric cardiac surgery with cardiopulmonary bypass (CPB). Enrollment will continue with a maximum of 350 subjects until 30 cases of AKI (stage 2 and 3) are reached.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Test fresh urine samples by NephroCheck | up to one year
  Urine samples for [TIMP-2]*[IGFBP7] measurements will be taken from each subject included in the study during the first 48 hours following cardiopulmonary bypass initiation according to the following schedule:
  * baseline before initiation of cardiopulmonary bypass (CPB, 0h).
  * - 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 48 hours after initiation of CPB

SECONDARY OUTCOMES:
Test serum creatinine and urea concentration to report AKI according KDIGO guideline | up to one year
  Blood samples for serum creatinine and urea concentration measurement will be taken from each subject included in the study during the first 48 hours following cardiopulmonary bypass initiation according to the following schedule:
  * baseline before initiation of cardiopulmonary bypass (CPB, 0 hours).
  * 12 hours, 24 hours, 48 hours, 60 hours after initiation of CPB

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jefferies JL, Devarajan P. Early detection of acute kidney injury after pediatric cardiac surgery. Prog Pediatr Cardiol. 2016 Jun;41:9-16. doi: 10.1016/j.ppedcard.2016.01.011. PMID 27429538
- [Result] Li S, Krawczeski CD, Zappitelli M, Devarajan P, Thiessen-Philbrook H, Coca SG, Kim RW, Parikh CR; TRIBE-AKI Consortium. Incidence, risk factors, and outcomes of acute kidney injury after pediatric cardiac surgery: a prospective multicenter study. Crit Care Med. 2011 Jun;39(6):1493-9. doi: 10.1097/CCM.0b013e31821201d3. PMID 21336114
- [Result] Morgan CJ, Zappitelli M, Robertson CM, Alton GY, Sauve RS, Joffe AR, Ross DB, Rebeyka IM; Western Canadian Complex Pediatric Therapies Follow-Up Group. Risk factors for and outcomes of acute kidney injury in neonates undergoing complex cardiac surgery. J Pediatr. 2013 Jan;162(1):120-7.e1. doi: 10.1016/j.jpeds.2012.06.054. Epub 2012 Aug 9. PMID 22878115
- [Derived] Tao Y, Heskia F, Zhang M, Qin R, Kang B, Chen L, Wu F, Huang J, Brengel-Pesce K, Chen H, Mo X, Liang J, Wang W, Xu Z. Evaluation of acute kidney injury by urinary tissue inhibitor metalloproteinases-2 and insulin-like growth factor-binding protein 7 after pediatric cardiac surgery. Pediatr Nephrol. 2022 Nov;37(11):2743-2753. doi: 10.1007/s00467-022-05477-6. Epub 2022 Feb 24. PMID 35211796